CLINICAL TRIAL: NCT04961138
Title: Pre-operative Neoadjuvant Therapy Combined With Surgery for Treating Stage III Hepatocellular Carcinoma: an Open, Random, Multicenter, Prospective Study
Brief Title: Pre-operative Neoadjuvant Therapy Combined With Surgery for Treating Stage III Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-01
Record Dates: First submitted 2019-10-16; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Hepatocellular Carcinoma Stage III
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Embolization, Therapeutic; lenvatinib; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant group (Experimental)
  Interventions: Procedure: Transhepatic Arterial Chemotherapy And Embolization (TACE)
- Surgery group (Active Comparator)
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Transhepatic Arterial Chemotherapy And Embolization (TACE) — Receiving TACE and lenvatinib before surgery.
  Other Names: lenvatinib
  Arms: Neoadjuvant group
Procedure: Surgery — Removing tumor by surgery.
  Arms: Surgery group

SUMMARY:
The purpose of present study is to evaluate whether per-operative neoadjuvant therapy combined with surgery could improve the 1-year disease-free survival of stage III hepatocellular carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old, both gender
* Confirmed diagnosis of stage III hepatocellular carcinoma(HCC)
* Fulfill the criteria of surgery
* No other severe comorbidity
* Eastern Cooperative Oncology Group score(ECOG) 0-2
* Expected survival > 3months
* Informed consent obtained.

Exclusion Criteria:

* Received chemoradiotherapy or other antineoplastic drugs
* Severe cirrhosis with Child-Pugh score >10
* Total bilirubin > 1.5 times upper limit, AST or ALT > 2times upper limit, indocyanine green retention rate after 15 min(ICG15) >=40%;
* Not fulfill the surgery criteria
* Received major surgery within 1month
* History of other tumor
* Participate other clinical trial within 1month
* Drug or alcohol abuse, AIDS
* Uncontrollable epileptic seizure or cognitive disorder
* Severe allergy
* Other unsuitable conditions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
1-year disease free survival | 1 year

SECONDARY OUTCOMES:
1-year overall survival | 1 year
Rate of R0 resection | 1 week
objective response rate | up to 2 months

IPD SHARING:
Plan to Share IPD: Undecided